#### NCT02780115

**Study ID**: 199201-010

**Title:** A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety, Efficacy, and Pharmacokinetics of the Fixed Combination of AGN-199201 and AGN-190584 in Patients With Presbyopia

Statistical Analysis Plan Amendment 2 Date: 15Dec2017

#### 1. Title Page

#### STATISTICAL ANALYSIS PLAN

A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety, Efficacy, and Pharmacokinetics of the Fixed Combination of AGN-199201 and AGN-190584 in Patients With Presbyopia

Amendment 2.0: 2017-12-15

Study Number: 199201-010

Development Phase: 2

Product Name: AGN-199201 (oxymetazoline hydrochloride

ophthalmic solution) and AGN-190584 (pilocarpine

hydrochloride ophthalmic solution)

Study Statistician:

Sponsor: Allergan PLC

2525 Dupont Drive, Irvine, California USA 92612

+1-714-246-4500

This document is the property of Allergan PLC and may not, in full or part, be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan PLC.

# 2. Table of Contents

| 1. | Title | Page | | 1 |
|---|---|---|---|---|
| 2. | Tabl | e of Cor | ntents | 2 |
| | 2.1 | List of | Tables | 3 |
| | 2.2 | | Figures | |
| 3. | List | | eviations and Definition of Terms | |
| 4. | Intro | duction | | 8 |
| | 4.1 | | Design Summary | |
| | 4.2 | _ | Objectives | |
| | 4.3 | _ | ule of Activities | |
| 5 | | | lethodology and Study Endpoints | |
| 5. | | | | |
| | 5.1 | Statist | ical Methods Planned in the Protocol and Determination of Sample Size | |
| | | 5.1.1 | Statistical and Analytical Plans | |
| | | | 5.1.1.1 Common Conventions | |
| | | | 5.1.1.2 Demographics | |
| | | | 5.1.1.3 Efficacy Analyses | |
| | | | 5.1.1.4 Safety Analyses | 30 |
| | | | | 20 |
| | | <i>5</i> 1 0 | 5.1.1.7 Interim Analyses | |
| | 5.0 | 5.1.2 | Determination of Sample Size | |
| | 5.2 | | es in the Conduct of the Study or Planned Analyses | |
| | | 5.2.1 | Changes in the Conduct of the Study | |
| | D ( | 5.2.2 | Changes to Analyses Prior to Database Lock | |
| 6. | Data | i Handiii | ng and Analysis Conventions | 39 |
| | 6.1 | Study | Treatment Conventions | 39 |
| | | 6.1.1 | Analysis Days | 39 |
| | | 6.1.2 | Missing/Incomplete Treatment End Date | 40 |
| | 6.2 | Analys | sis Visit Windows | 40 |
| | | 6.2.1 | Safety | 40 |
| | 6.3 | Site Po | poling | 41 |
| | 6.4 | Missir | ng/Incomplete Date Conventions | 41 |
| | | 6.4.1 | Missing/Incomplete AE Start Date | 41 |
| | | 6.4.2 | Missing/Incomplete Medication Start Date | 41 |

| | 6.4.3 Missing/Incomplete AE/Medication End Date | 42 |
|------------|--------------------------------------------------|----|
| 6.5 | Efficacy Endpoint Conventions | 42 |
| 6.6 | Safety Endpoint Conventions. | 42 |
| | 6.6.1 Adverse Events | 42 |
| | 6.6.1.1 Missing Intensity or Relationship | |
| | 6.6.1.2 Possible Distant Spread of Toxin (PDSOT) | |
| | 6.6.1.3 AE Group of Interest | 42 |
| - <b>-</b> | 6.6.4 Electrocardiograms | |
| 6.7 | Imputed Value Listing Conventions | |
| 6.8 | Analysis Plan Amendment 1 Summary | |
| 6.9 | Analysis Plan Amendment 2 Summary | 44 |
| 2.1 | List of Tables | |
| Table 3-1 | Abbreviations and Definitions of Terms. | 6 |
| Table 4-1 | Study Treatment Group | 9 |
| Table 4-2 | Study Objectives | 9 |
| Table 5-1 | Analysis Populations | 20 |
| Table 5-2 | Statistical Methodology | 21 |
| Table 5-3 | Missing Data Handling by Endpoint Type | 22 |
| Table 5-4 | Analysis Population Summaries | 22 |
| Table 5-5 | Subject Disposition Summaries | 23 |

| Table 5-6 | Protocol Deviation Summary | 23 |
|------------|-----------------------------------------------------------|----|
| Table 5-7 | Demographic Summaries | 23 |
| Table 5-8 | Baseline Characteristics Summaries | 23 |
| Table 5-9 | Medical History Summary | 24 |
| Table 5-10 | Ophthalmic History and Ophthalmic Surgery History Summary | 24 |
| Table 5-11 | Medication Summaries | 25 |
| Table 5-14 | Mesopic, High Contrast UNVA | 26 |
| Table 5-24 | AE Terms | 31 |
| Table 5-25 | AE Summaries | 31 |

| e 6-4 Imputation Scenarios | |
|---|---|
| e 6-4 Imputation Scenarios | |
| e 6-4 Imputation Scenarios | |
| 6-4 Imputation Scenarios | |
| 5-4 Imputation Scenarios | |
| 5-4 Imputation Scenarios | |
| -4 Imputation Scenarios | |
| -4 Imputation Scenarios | |
| Initial Imputed Date Algorithm | Analysis Day Definitions |
| Initial Imputed Date Algorithm | |
| Initial Imputed Date Algorithm | |
| | Imputation Scenarios |
| Mississ AT Intercent Deletional in Insertation Alexandres | Initial Imputed Date Algorithm |
| Missing AE Intensity and Relationship Imputation Algorithms | Missing AE Intensity and Relationship Imputation Algorithms |
| | List of Figures |
| List of Figures | |

## 3. List of Abbreviations and Definition of Terms

Table 3-1 Abbreviations and Definitions of Terms

| Abbreviation/Term | Definition |
|---|---|
| AE | adverse event |
| AGN | Allergan |
| ANCOVA | analysis of covariance |
| ANOVA | analysis of variance |
| ATC | Anatomical Therapeutic Chemical |
| CFB | change from baseline |
| CMH | Cochran-Mantel-Haenszel |
| DCNVA | distance corrected near visual acuity |
| eCRF | electronic case report form |
| GCP | Good Clinical Practice |
| ICH | International Conference on Harmonisation |
| IOP | intraocular pressure |
| IxRS | interactive response system |
| LOCF | last observation carried forward |
| LS | least squares |
| MedDRA | Medication Dictionary for Regulatory Activities |
| mITT | modified intent-to-treat |
| N | number of patients |
| N/A | not applicable |
| NEI | national eye institute |
| NVPT | near vision presbyopia task |
| OC | observed cases |
| OCT | optical coherence tomography |
| OU | both eyes |
| PCS | potentially clinically significant |
| PICO PRO | presbyopia impact and coping questionnaire patient-reported outcome |
| PO | primary objective |
| PP | per-protocol |
| PPSQ PRO | presbyopia patient satisfaction questionnaire patient-reported outcome |
| PRO | patient-reported outcome |
| PT | preferred term |
| QD | once daily |
| SAE | serious adverse event |
| SADE | serious adverse device effect |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SE | standard error |
| SO | secondary objective |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| UDVA | uncorrected distance vision acuity |
| UNVA | uncorrected near vision acuity |
| VAS | visual analog scale |
| ı | - |

| Abbreviation/Term | Definition |
|-------------------|---------------------------|
| WHO | World Health Organization |

#### 4. Introduction

This statistical analysis plan (SAP) details comprehensive, technical specifications of the statistical analyses of the efficacy, safety data and health outcomes outlined and/or specified in the final protocol of Study 199201-010 (version dated 2015-10-28) and the most recent amendment (version 3 dated 2016-08-18). Specifications of tables, figures, and data listings are contained in a separate document. The SAP for pharmacokinetic/pharmacodynamic and/or health economics and outcomes research data will be prepared separately. This document is organized into 3 main sections:

- 1. Study overview
- 2. Statistical Methodology and Study Endpoints
- 3. Data Handling and Analysis Conventions

#### 4.1 Study Design Summary

This multicenter, double-masked, randomized, parallel-group, vehicle-controlled study will be a controlled comparison of fixed combinations of AGN-199201 and AGN-190584 at different concentrations to vehicle dosed in both eyes (OU), and the fixed combination of AGN-199201 and AGN-190584 dosed in OU or in the nondominant eye only. Study medication will be administered once daily (QD) in the morning. During office visits 1 through 5, study medication will be administered at hour 0 (8 AM  $\pm$  1 hour). Following the treatment period, all patients will be seen for a  $14 \pm 2$ -day follow-up period as shown in Figure 1. The study duration will be 38 to 65 days per patient.



Table 4-1 Study Treatment Group

| Treatment Group | AGN-199201 (%) | AGN-190584 (%) | Dosing |
|-----------------|-----------------|-----------------|-----------------|
| 1 | Vehicle control | Vehicle control | OU |
| 2 | | | OU |
| 3 | | | OU |
| 4 | | | OU |
| 5 <sup>a</sup> | | | Nondominant eye |

OU = both eyes

# 4.2 Study Objectives

Each study primary objective (PO), and secondary objective (SO) are presented below:

Table 4-2 Study Objectives

| · |
|---|
| Objectives |
| PO To evaluate the safety, efficacy, and tolerability of fixed combinations of AGN-199201 and AGN-190584 over a 42-day observation period when administered bilaterally, once daily (QD) for 28 days in patients with presbyopia |
| SO1 To compare the safety, efficacy, and tolerability of a fixed combination of AGN-199201 and AGN-190584 when administered monocularly to the nondominant eye versus bilaterally over a 42-day observation period with QD dosing for the first 28 days in patients with presbyopia |
| SO2 To assess the systemic pharmacokinetics of AGN-199201 and AGN-190584 following single and multiple (QD for 28 days) ophthalmic administrations as a fixed combination in 1 or both eyes (OU) |
| SO3 To evaluate the psychometric properties of the de novo patient-reported outcome (PRO) instruments developed for this program, including the near vision presbyopia performance tasks and task-based questionnaire under mesopic and photopic conditions, the presbyopia patient satisfaction questionnaire, and the presbyopia impact and coping questionnaire |

PO = primary objective, SO1 = first secondary objective, SO2 = second secondary objective, SO3 = third secondary objective

<sup>&</sup>lt;sup>a</sup> Dominant eye dosed with vehicle





















#### 5. Statistical Methodology and Study Endpoints

# 5.1 Statistical Methods Planned in the Protocol and Determination of Sample Size

This statistical analysis plan (SAP) will be approved prior to database lock. The SAP expands the statistical section of the protocol and contains a detailed description of methods to analyze data collected in the study. The text portion of the SAP will be included in the CSR report as Appendix 16.1.9.

#### 5.1.1 Statistical and Analytical Plans

Statistical analyses will be conducted using

#### **5.1.1.1** Common Conventions

#### 5.1.1.1.1 Analysis Populations

The analysis populations will consist of patients as defined below: See Table 5-1.

Table 5-1 Analysis Populations

| Population | Population Definition | |
|---|---|---|
| Screened | ened All screened patients who sign informed consent | |
| Modified Intent-to- | All randomized patients with a baseline and at least 1 post | Randomized assignment |
| Treat (mITT) | baseline assessment of mesopic, high contrast, UNVA and will | _ |
| be analyzed as randomized | | |
| Safety | All patients who received $\geq 1$ administration of study treatment | Actual received |
| | and will be analyzed as treated | |

The efficacy variables will be analyzed using the mITT population. All safety measures will be analyzed using the safety population.

#### **5.1.1.1.2** Study Treatments

The following treatment groups are defined for this study, also presented in Table 4-1, as group 1, 2, 3, 4 and 5:

- Group 1: Vehicle Control, OU
- Group 2: Fixed combination AGN-199201 and AGN-190584 ), OU
- Group 3: Fixed combination AGN-199201 and AGN-190584 OU
- Group 4: Fixed combination AGN-199201 and AGN-190584 , OU
- Group 5: Fixed combination AGN-199201 and AGN-190584 Non-dominant eye and vehicle to the dominant eye

#### 5.1.1.1.3 Statistical Methodology

The methodologies defined below apply as specified to individual endpoints defined in this SAP. When indicated, 95% two-sided confidence intervals and two-sided p-values will be presented. Individual endpoint analyses may specify exceptions (additions or deletions) to these general definitions.

Table 5-2 Statistical Methodology

| Methodology | | Description |
|---|---|---|
| M1 | Categorical | Number of patients in individual categories |
| | counts | o Patients with ≥ 1 qualifying event counted once per individual category |
| M2 | Categorical descriptives | <ul> <li>Number and percentage of patients in individual categories <ul> <li>Patients with ≥ 1 qualifying event counted once per individual category</li> </ul> </li> <li>(Optional) N included if percentage denominator ≠ number of patients in the population (standard percentage denominator).</li> </ul> |
| M3 | PCS<br>descriptives | <ul> <li>Number and percentage of patients meeting potentially clinically significant (PCS) criteria <ul> <li>Patients with ≥ 1 qualifying event counted once per PCS category</li> </ul> </li> <li>Percentage denominator = number of patients with non-missing baseline and &gt;=1 non-missing postbaseline assessment</li> <li>Unevaluable assessments considered missing</li> </ul> |
| M4 | Continuous descriptives | <ul> <li>N included, mean, standard deviation (SD), median, minimum, maximum</li> <li>N included = patients with non-missing value</li> </ul> |
| M5 | CFB descriptives | <ul> <li>Continuous descriptives for baseline, postbaseline, and change from baseline (CFB) values</li> <li>N included = patients with non-missing values at both baseline and the specified postbaseline analysis visit</li> </ul> |
| M6 | CFB<br>ANCOVA | <ul> <li>Continuous descriptives and standard error (SE) for baseline, postbaseline, and CFB values</li> <li>Estimates derived from mixed model for CFB value controlling for treatment group and covariates (baseline UNVA severity, iris color and age group) <ul> <li>Least squares (LS) means and standard errors</li> <li>P-values and confidence intervals from contrast t-test comparing active AGN-199201 treatment groups vs AGN-199201 vehicle</li> </ul> </li> <li>N included = patients with non-missing values at both baseline and the postbaseline analysis visit</li> </ul> |
| M7 | CFB figure | <ul> <li>Plot of CFB LS means and SE bars for each treatment group</li> </ul> |
| M8 | Responder | <ul> <li>Categorical descriptives for responders and nonresponders <ul> <li>Nonresponders include:</li> <li>Patients who do not meet responder criteria</li> </ul> </li> <li>CMH test comparing active AGN-199201 treatment groups vs AGN-199201 vehicle</li> </ul> |

ANCOVA = analysis of covariance; N = number of patients. CMH = Cochran-Mantel-Haenszel Raw and derived data listings will be provided, and will be fully defined in the table, figure, and data listing specification document.

## **5.1.1.1.4 Missing Data**

There will be no imputation of missing data for all analyses.

| Table 5-3 | Missing Data Handling by Endpoint Type | e |
|-----------|----------------------------------------|---|

| <b>Endpoint type</b> | Timing | Missing Data Handling |
|---|---|---|
| Responder | Treatment Period | All patients included |
| | | Patients with no postbaseline values will be excluded |
| CFB ANCOVA | Treatment Period | <ul> <li>If missing covariates (including baseline if applicable) <ul> <li>Subject excluded</li> </ul> </li> <li>If missing average change from baseline UNVA letters: <ul> <li>Subject excluded</li> </ul> </li> </ul> |
| CFB Posebaseline | Treatment Period | <ul> <li>If missing value at the specified postbaseline analysis visit: <ul> <li>Available cases</li> <li>Subject excluded</li> </ul> </li> </ul> |

ANCOVA = analysis of covariance; CFB = change from baseline

#### **5.1.1.1.5 Site Pooling**

Data from all sites will be pooled for analysis.

#### **5.1.1.1.6 Other Common Conventions**

Ocular adverse events and other ocular evaluations will be summarized using eye as the experimental unit by treatment group. Nonocular adverse events and other nonocular assessments will be summarized using patient as the experimental unit by treatment group.

#### **5.1.1.2 Demographics**

#### 5.1.1.2.1 Analysis Populations

The distribution of patients within the analysis populations will be summarized as follows:

Table 5-4 Analysis Population Summaries

| Population | Description | Timing | Methodology |
|---|---|---|---|
| Screened Population | Distribution overall and within | Screening Period | Categorical counts |
| | countries/regions/sites in total | | |
| mITT and Safety | Distribution overall and within | Treatment Period | Categorical counts |
| populations | countries/regions/sites in total and by | | |
| | treatment group | | |

#### **5.1.1.2.2** Participant Disposition

Subject disposition encompasses the distribution of patients who enter, complete, and discontinue each specified analysis period, along with electric case report form (eCRF)-reported discontinuation reasons from each respective analysis period. Subject disposition will be summarized as follows:

Table 5-5 Subject Disposition Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Screening disposition | Distribution in the Screened | Screening Period | Categorical descriptive |
| | Population in total | | |
| Study disposition | Distribution in the mITT Population | Treatment Period | Categorical descriptive |
| | in total and by treatment group | | |

mITT = modified intent-to-treat

#### 5.1.1.2.3 Protocol Deviations

Protocol deviations will be defined in a separate document, including importance classification. Protocol deviations will be summarized as follows:

Table 5-6 Protocol Deviation Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Important protocol | Distribution in the mITT Population | Treatment Period | Categorical descriptive |
| deviations | in total and by treatment group | | |

#### 5.1.1.2.4 Demographics

Demographics will be summarized for the Screened Population, and in total and by treatment group for the mITT and Safety populations, as follows:

Table 5-7 Demographic Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Age | Age (years) relative to informed consent | Informed consent | Continuous |
| | date | | descriptives |
| Age group | • ≤ 50 years | Informed consent | Categorical |
| | • > 50 years | | descriptives |
| Sex, race, and | eCRF categories | Screening Period | Categorical |
| ethnicity | Race group | | descriptives |
| | o White | | |
| | o Non-white | | |
| | Ethnicity | | |
| | o Hispanic | | |
| | <ul> <li>Non-hispanic</li> </ul> | | |

#### **5.1.1.2.5** Baseline Characteristics

Baseline characteristics will be summarized in total and by treatment group for the mITT and Safety populations as follows:

 Table 5-8
 Baseline Characteristics Summaries

| Parameter | Description | Timing | Methodology |
|--------------------------|-------------|----------------------|-------------|
| Baseline characteristics | Iris color | Latest assessment in | Categorical |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| | | Screening Period or | descriptives |
| | | Pretreament Period | |
| Randomization strata | • UNVA severity at baseline (≤ 20/80 and > 20/80) | Randomization date | Categorical descriptives |
| Baseline efficacy | <ul> <li>Mesopic pupil diameter with<br/>Grand Seiko sites vs without<br/>Grand Seiko sites</li> <li>UNVA severity at baseline<br/>with Grand Seiko sites vs<br/>without Grand Seiko sites</li> </ul> | Randomization date | Continuous<br>descriptives |

## 5.1.1.2.6 Medical History

Medical history, encompassing abnormalities and surgeries reported as occurring before the Screening Visit, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 19.0 or newer. Unique patients who report medical history events will be summarized by MedDRA system organ class (SOC) and preferred term (PT) by treatment group for the Safety Population as follows:

Table 5-9 Medical History Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Medical and surgical | Abnormalities and surgeries occurring | Screening Period | Categorical |
| history | before the Screening Visit | | descriptive |

SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose group.

## 5.1.1.2.7 Ophthalmic History and Ophthalmic Surgical History

Ophthalmic history, encompassing abnormalities and ophthalmic surgeries reported as occurring before the Screening Visit, will be coded using MedDRA, version 19.0 or newer. Unique patients who report ophthalmic history events will be summarized by MedDRA SOC and PT by treatment group for the Safety Population as follows:

Table 5-10 Ophthalmic History and Ophthalmic Surgery History Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Ophthalmic history and | Abnormalities and surgeries occurring | Screening Period | Categorical |
| ophthalmic surgery | before the Screening Visit | | descriptive |
| history | | | |

SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose group.

#### 5.1.1.2.8 Prior and Concomitant Medications

Medications will be listed for the Safety Population as follows:

Medications will be coded using the World Health Organization (WHO) Drug Dictionary, version 14.0 or newer. Unique patients who reported medications will be summarized by

Anatomical Therapeutic Chemical (ATC) 4 class and PT by treatment group for the Safety Population as follows:

**Table 5-11 Medication Summaries** 

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Prior medications | Medications taken $\geq 1$ time before | Screening Period, | Categorical |
| | the study treatment start date, | Pretreament Period | descriptives |
| | regardless of medication end date | | |
| Concomitant | Medications taken $\geq 1$ time on or after the | Treatment Period, | Categorical |
| medications | study treatment start date, regardless of | Follow-up Period | descriptives |
| | medication start date | | _ |
| | <ul> <li>Medications starting 1 day after</li> </ul> | | |
| | treatment end date will be listed | | |
| | but excluded from analysis | | |

ATC4 classes will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose group.

## **5.1.1.3** Efficacy Analyses

Efficacy analyses will be based on the mITT Population.

The following efficacy assessments are defined:



Baseline assessments for applicable efficacy endpoints defined as follows:

Table 5-13 Efficacy Endpoint Baseline Definitions

| Endpoint | Description | Timing |
|---|---|---|
| Mesopic, high contrast UNVA | Non-missing measurements at Day 1 Hour 0 • Patients with no Day 1 Hour 0 measurement will be excluded from CFB analyses¹ | Day 1 Hour 0 |
| - | | |
| - | | |

## 5.1.1.3.1 Study Success Criteria

There will be no adjustment of type 1 error rate for the multiple tests. There will be no imputation of missing data for all analyses.

## 5.1.1.3.2 Mesopic, High Contrast UNVA

Mesopic, high contrast UNVA endpoints will be summarized by treatment group for mITT Population.

Table 5-14 Mesopic, High Contrast UNVA

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Average change from | Average change from baseline in UNVA lines in the | Treatment | CFB |
| baseline in UNVA | nondominant eye at day 28. | Period Day | ANCOVA <sup>1</sup> |
| letters (Primary efficacy | | 28 | CFB figure |
| variable) | | | |







#### 5.1.1.4.2 Adverse Events

The following adverse event (AE) terms are defined:

Table 5-24 AE Terms

| Term | Description |
|---|---|
| Treatment- | An event that initially occurs or increases in intensity on or after the treatment start date, where: |
| emergent | <ul> <li>Treatment start date ≤ event start date ≤ treatment end date + 30</li> </ul> |
| On-therapy | An event where: |
| | • Treatment start date ≤ event start date ≤ treatment end date + 30 |

AEs, encompassing abnormalities and surgeries reported as occurring after the Screening Visit, will be coded using MedDRA version 19.0 or newer. Unique patients reporting AEs in the following AE categories will be summarized by treatment group and overall for the Safety Population as follows:

Table 5-25 AE Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Overall summary | Overall summary only for the following categories: • Treatment-emergent AEs (TEAEs) • Treatment-related TEAEs • Study-procedure-related TEAEs • On-therapy serious adverse events (SAEs) • On-therapy fatal SAEs • AEs leading to discontinuation | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| TEAEs | Overall summary and by SOC and PT | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Ocular TEAEs | Summary by SOC and PT for ocular TEAEs dominant eye nondominant eye | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Non-ocular TEAEs | Summary by SOC and PT for non-ocular TEAEs | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Common TEAEs | Summary by PT • Includes TEAEs occurring in ≥ 5.0% of patients in any treatment group | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Common Ocular<br>TEAEs | Summary by PT for common ocular TEAEs dominant eye | Treatment Period,<br>Follow-up Period | Categorical descriptives |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| | nondominant eye | | <u> </u> |
| Common Non-ocular<br>TEAEs | Summary by PT for common non-ocular TEAEs | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| TEAEs by intensity | Overall summary and by SOC, PT, and intensity • Patients categorized overall and | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| | within each SOC and PT for the most intense occurrence | | |
| Ocular TEAEs by intensity | Overall summary and by SOC, PT, and intensity for ocular TEAEs • Patients categorized overall and within each SOC and PT for the most intense occurrence dominant eye nondominant eye | Treatment Period,<br>Follow-up Period | Categorical<br>descriptives |
| Non-ocular TEAEs by intensity | Overall summary and by SOC, PT, and intensity for non-ocular TEAEs • Patients categorized overall and within each SOC and PT for the most intense occurrence | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Treatment-related | Overall summary and by PT | Treatment Period, | Categorical |
| TEAEs | | Follow-up Period | descriptives |
| Ocular Treatment-related TEAEs | Overall summary and by PT for ocular TEAEs dominant eye nondominant eye | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Non-ocular Treatment- | Overall summary and by PT for non-ocular | Treatment Period, | Categorical |
| related TEAEs | TEAEs | Follow-up Period | descriptives |
| Study-procedure-related TEAEs | Overall summary and by PT | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Ocular Study-<br>procedure-related<br>TEAEs | Overall summary and by PT for ocular TEAEs dominant eye nondominant eye | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| Non-ocular Study-<br>procedure-related<br>TEAEs | Overall summary and by PT for non-ocular TEAEs | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| On-therapy SAEs <sup>1</sup> | Overall summary and by PT | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| On-therapy ocular<br>SAEs | Overall summary and by PT for ocular SAEs dominant eye nondominant eye | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| On-therapy non-ocular | Overall summary and by PT for non-ocular | Treatment Period, | Categorical |
| SAEs | SAEs | Follow-up Period | descriptives |
| On-therapy fatal SAEs <sup>1</sup> | Overall summary and by PT | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| On-therapy fatal ocular SAEs | Overall summary and by PT for ocular fatal SAEs dominant eye | Treatment Period,<br>Follow-up Period | Categorical descriptives |
| | nondominant eye | | |
| On-therapy fatal<br>non-ocular SAEs | Overall summary and by PT for non-ocular fatal SAEs | Treatment Period,<br>Follow-up Period | Categorical descriptives |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| AEs leading to study | Overall summary and by PT | Treatment Period, | Categorical |
| discontinuation <sup>1</sup> | | Follow-up Period | descriptives |
| Ocular AEs leading to | Overall summary and by PT for ocular | Treatment Period, | Categorical |
| study discontinuation | AEs leading to discontinuation | Follow-up Period | descriptives |
| | dominant eye | _ | _ |
| | nondominant eye | | |
| Non-ocularAEs leading | Overall summary and by PT for non-ocular | Treatment Period, | Categorical |
| to study discontinuation | AEs leading to discontinuation | Follow-up Period | descriptives |

<sup>&</sup>lt;sup>1</sup> Patients who report ≥ 1 AE in the AE category and all AEs for those patients will be listed. SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose group.







## 5.1.1.7 Interim Analyses

Not applicable

## **5.1.2 Determination of Sample Size**

A sample size of approximately 150 patients will be randomized in a 1:1:1:1:1 ratio into 1 of the 5 study groups. Approximately two-thirds of the enrolled patients will be younger patients ( $\leq$  50 years old), and approximately one-third of the enrolled patients will be older patients (> 50 years old).

From the Study 199201-007 results, the treatment effect for the younger patients was on average 1.98 lines of change in mesopic, high contrast UNVA, with standard deviations for active and

vehicle of 1.12 and 1.01, respectively. For older patients, the treatment effect was on average 0.72 lines of change in mesopic, high contrast UNVA, with standard deviations for active and vehicle of 1.87 and 1.15, respectively. The treatment effect for the younger patients was on average 1.02 lines of change in photopic, high contrast UNVA, with standard deviations for active and vehicle of 1.42 and 0.67, respectively. For older patients, the treatment effect was on average 0.27 lines of change in photopic, high contrast UNVA, with standard deviations for active and vehicle of 1.10 and 0.93, respectively.

Accounting for a 12.5% dropout rate, 26 patients per treatment group will provide 99% power to observe a difference between an active group and the vehicle group for lines of change from baseline in mesopic, high contrast UNVA, and 68% power for lines of change from baseline in photopic, high contrast UNVA, with a type I error of 0.05

#### 5.2 Changes in the Conduct of the Study or Planned Analyses

#### 5.2.1 Changes in the Conduct of the Study

Not applicable

#### **5.2.2** Changes to Analyses Prior to Database Lock

The term of 'average change from baseline in UNVA letters' instead of 'weighted average change from baseline in UNVA letters' will be used since weighted average concept only applies when missing mid-timepoint values are imputed. UNVA responder analyses with at least a 2-line improvement in mesopic, high contrast UNVA from baseline at a majority of postdose timepoints (6 or more) in the nondominant eye will be added.

Subgroup analyses by gender, race and ethnicity will not be performed.

#### 6. Data Handling and Analysis Conventions

## **6.1 Study Treatment Conventions**

#### 6.1.1 Analysis Days

Treatment is defined as follows:

Table 6-1 Analysis Day Definitions

| Term | Description |
|---------------|--------------------------------------------------|
| Treatment Day | Relative to treatment start date |
| | If analysis date ≥ treatment start date: |
| | • Day = analysis date – treatment start date + 1 |
| | o Day 1 = treatment start date |
| | · |

## **6.1.2 Missing/Incomplete Treatment End Date**

If the investigator is unable to provide the treatment end date, treatment end date will be imputed as the last available dosing record date/last available efficacy assessment date





## 6.3 Site Pooling

Data from all sites will be pooled for analysis.

## 6.4 Missing/Incomplete Date Conventions

Dates may be imputed with year, month, and day values under certain scenarios:

Table 6-4 Imputation Scenarios

| | Complete | | | |
|----------|----------|-------|-----|-----------------|
| Scenario | Year | Month | Day | Imputable |
| 1 | Yes | Yes | Yes | Complete |
| 2 | Yes | Yes | _ | Yes |
| 3 | Yes | _ | Yes | No <sup>1</sup> |
| 4 | Yes | _ | _ | Yes |
| 5 | _ | Yes | Yes | No <sup>1</sup> |
| 6 | _ | Yes | _ | No <sup>1</sup> |
| 7 | _ | _ | Yes | No <sup>1</sup> |
| 8 | _ | _ | _ | Yes |

<sup>&</sup>lt;sup>1</sup> Not allowed per database design.

Dates will be imputed initially toward a specified target date for imputable scenarios 2, 4, and 8, and adjusted against the latest reasonable dates. The initial imputed date is determined by the following algorithm:

Table 6-5 Initial Imputed Date Algorithm

| Available Year | | Available Month (MM) | | |
|---|---|---|---|---|
| (YYYY) | Missing | < Target Month = Target Month > Target Month | | |
| Missing | Target Date | | _ | |
| < Target Year | YYYY-12-31 | | YYYY-MM-LD | |
| = Target Year | Target Date | YYYY-MM-LD | Target Date | YYYY-MM-01 |
| > Target Year | YYYY-01-01 | | YYYY-MM-01 | |

YYYY = available start date year; MM = available start date month; LD = last day of the month.

## 6.4.1 Missing/Incomplete AE Start Date

AE start dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = Treatment start date
- Complete end date

## **6.4.2 Missing/Incomplete Medication Start Date**

Medication start dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = Treatment start date -1
- Complete end date

#### 6.4.3 Missing/Incomplete AE/Medication End Date

AE and medication end dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = Treatment end date + 30
- Death date

## 6.5 Efficacy Endpoint Conventions

Not applicable

#### **6.6** Safety Endpoint Conventions

#### **6.6.1** Adverse Events

#### 6.6.1.1 Missing Intensity or Relationship

If the investigator is unable to provide the actual values, the following imputations will be applied:

Table 6-6 Missing AE Intensity and Relationship Imputation Algorithms

| Missing Value | Imputation | Timing |
|---------------|--------------|---------------------------------------|
| Intensity | Mild | Screening Period, Pretreatment Period |
| | Severe | Treatment Period |
| Relationship | <del>_</del> | Screening Period, Pretreatment Period |
| | Related | Treatment Period |

# **6.6.1.2** Possible Distant Spread of Toxin (PDSOT)

Not applicable

### 6.6.1.3 **AE Group of Interest**

Not applicable



#### 6.6.4 Electrocardiograms

Not applicable

#### 6.7 Imputed Value Listing Conventions

In general, listings will present the actual partial or missing values rather than the imputed values that may be used in endpoint derivation. In instances where imputed values will be presented, imputed values will be flagged. Actual rules will be fully defined in the table, figure, and data listing specification document.

#### 6.8 Analysis Plan Amendment 1 Summary

Following is a summary of content-oriented changes that were made to each section of the protocol, and a brief rationale for these changes. Minor editorial and document formatting revisions have not been summarized.



| Section | Revision | Rationale |
|---------|-------------------------------|-----------|
| | timepoints (6 or more) in the | |
| | nondominant eye will be | |
| | added | |

#### 6.9 Analysis Plan Amendment 2 Summary

Following is a summary of content-oriented changes that were made to each section of the protocol, and a brief rationale for these changes. Minor editorial and document formatting revisions have not been summarized.



# **ALLERGAN**

# 199201-010 Statistical Analysis Plan

| Date (DD/MMM/YYYY)/Time (PT) | Signed by: | Justification |
|------------------------------|------------|---------------|